CLINICAL TRIAL: NCT03625687
Title: Pan-genotypic Direct Acting Antiviral Therapy in Donor HCV-positive to Recipient HCV-negative Lung Transplant
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funding, transitioned to standard of care
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Raymond Chung, Director of Hepatology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2018P001697
Record Dates: First submitted 2018-07-30; First posted 2018-08-10 (Actual); Results first posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Respiratory Failure; Hepatitis C
Keywords: Lung disease; Lung Transplant; HCV; Hepatitis C
MeSH Terms: conditions — Respiratory Insufficiency; Hepatitis C; Lung Diseases | interventions — glecaprevir and pibrentasvir; sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with Direct Acting Antiviral for HCV (Experimental): 8 weeks of treatment with HCV Direct Acting Antiviral tablet (Mavyret or Epclusa)
  Interventions: Drug: Clinically prescribed direct acting antiviral (Mavyret or Epclusa) HCV treatment for 8 weeks

INTERVENTIONS:
Drug: Clinically prescribed direct acting antiviral (Mavyret or Epclusa) HCV treatment for 8 weeks — 8 weeks of direct acting antiviral treatment based on clinical indication (either Mavyret or Epclusa)
  Other Names: DAA treatment; Mavyret; Epclusa

SUMMARY:
This is a proof of concept, single center study for the donation of HCV-positive lungs to HCV negative recipient patients, with preemptive, interventional treatment with 8 weeks of commercially available DAA therapy to prevent HCV transmission upon transplantation.

DETAILED DESCRIPTION:
The goal of this study is to determine if preoperative dosing and sustained administration of pan-genotypic DAA therapy after lungs transplantation prevents the transmission of hepatitis C virus (HCV) infection from an HCVpositive donor lung to an HCV naïve recipient.

ELIGIBILITY:
Inclusion Criteria:

* Met MGH transplant center criteria, listed for lung transplant
* Able to sign informed consent

Exclusion Criteria:

* Pregnant or nursing (lactating) women
* HIV positivity
* Any contra-indication to lung transplantation per center protocol
* For study patients in whom Epclusa® therapy is being considered, exclusion criteria includes patients on the following p-glycoprotein inducers or moderate to potent CYP inducers that cannot stop therapy: carbamazepine, phenytoin, phenobarbital, oxcarbazepine, rifabutin, rifampin, rifapentine, St. John's wort.
* For study patients in whom MavyretTM therapy is being considered, exclusion criteria includes patients on the following medications who cannot stop therapy: carbamazepine, rifampin, St. John's wort, and ethinyl estradiol-containing oral contraceptives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond T Chung, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Anticipate to share coded data with collaborators
Supporting Information: Study Protocol
Time Frame: Anticipate data would be available to share within 6 months after the final patient completes the study.
Access Criteria: Coded data would be shared with collaborators who have received IRB approval to use the data and have been approved by the PI for their collaboration.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between February 2019 and December 2020.
Pre-assignment Details: 19 subjects received transplant with an HCV Ab positive organ. 3 of the 19 subjects received an HCV Ab positive/HCV RNA negation (NAT negative) transplant and did not irequire DAA therapy per protocol. 16 subjects received HCV Ab positive/HCV RNA positive (NAT positive) transplant and initiated DAA therapy.
Groups:
- Treatment With Direct Acting Antiviral for HCV: 8 weeks of treatment with HCV Direct Acting Antiviral tablet (Mavyret)
  Clinically prescribed direct acting antiviral (Mavyret) HCV treatment for 8 weeks: 8 weeks of direct acting antiviral treatment based on clinical indication (Mavyret)
Period: Overall Study
Arm/Group | Treatment With Direct Acting Antiviral for HCV
Started | 16
Completed | 15
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: Subjects receiving HCV RNA positive lung transplant and initiating treatment with DAA
Groups:
- Treatment With Direct Acting Antiviral for HCV: 8 weeks of treatment with HCV Direct Acting Antiviral tablet (Mavyret)
  Clinically prescribed direct acting antiviral (Mavyret) HCV treatment for 8 weeks: 8 weeks of direct acting antiviral treatment based on clinical indication (either Mavyret)
Arm/Group | Treatment With Direct Acting Antiviral for HCV
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants] — Age collected at time of consent.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 11
    >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16
Recipient HCV negative status at time of consent [Count of Participants; unit: Participants] | 16

OUTCOME MEASURES:

1. Primary Outcome: Undetectable Blood HCV RNA Level
Description: Negative HCV RNA by blood testing at 12 weeks after the last dose of treatment.
Time Frame: 12 weeks post last dose of treatment with DAA
Population: Number of subjects completing full course of treatment
Measure: Count of Participants; unit: Participants
Groups:
- Treatment With Direct Acting Antiviral for HCV: 8 weeks of treatment with HCV Direct Acting Antiviral tablet (Mavyret)
  Clinically prescribed direct acting antiviral HCV treatment for 8 weeks: 8 weeks of direct acting antiviral treatment based on clinical indication
Arm/Group | Treatment With Direct Acting Antiviral for HCV
Number analyzed (Participants) | 15
Participants | 15

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: Safety and tolerability of DAA therapy in the lung transplant recipient monitored by quantifying the number of treatment related adverese events per patient and evaluation clinically significant out of range lab results as compared to baseline/pretreatment values per patient
Time Frame: 8 weeks
Population: Number of participants receiving at least 1 dose of DAA treatment were included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Direct Acting Antiviral for HCV
Number analyzed (Participants) | 16
Participants | 0

3. Secondary Outcome: Tolerability (Based on Number of Adverse Events and Clinically Significant Laboratory Values)
Description: Tolerability of commercially available DAA therapy in the lung transplant patient will be monitored by quantifying the number of treatment related adverse events per patient and evaluating clinically significant laboratory results
Time Frame: 8 weeks
Population: Number of participants receiving at least one dose of DAA were included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Direct Acting Antiviral for HCV
Number analyzed (Participants) | 16
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of Direct Acting Antiviral Treatment initiation through last dose of therapy (8 week treatment period)
Description: Only treatment emergent adverse events were collected.
Groups:
- Treatment With Direct Acting Antiviral for HCV: Eight weeks of treatment with HCV Direct Acting Antiviral tablet (Mavyret or Epclusa)
  Clinically prescribed direct acting antiviral (Mavyret or Epclusa) HCV treatment for 8 weeks: 8 weeks of direct acting antiviral treatment based on clinical indication (either Mavyret or Epclusa)
Arm/Group | Treatment With Direct Acting Antiviral for HCV
All-Cause Mortality (participants affected / at risk) | 1/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

LIMITATIONS AND CAVEATS:
Study was terminated prior to completion and prior to meeting enrollment goal primarily due to lack of resources (staffing and funding) and transition of HCV-positive to HCV-negative lung transplants to standard of care. Full planned analysis was not completed due to enrollment number, however primary endpoint was assessed for all 16 subjects receiving treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/87/NCT03625687/Prot_SAP_000.pdf